CLINICAL TRIAL: NCT05904743
Title: INHALE-3: A 17-Week Randomized Trial and a 13-Week Extension, Evaluating the Efficacy and Safety of Inhaled Insulin (Afrezza) Combined With Insulin Degludec Versus Usual Care in Adults With Type 1 Diabetes
Brief Title: INHALE-3: Afrezza® Combined With Insulin Degludec Versus Usual Care in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-193
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Insulin; Inhaled; Afrezza; Technosphere; Adults; Degludec; Glucose sensors; Insulin pumps; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance; Respiratory Aspiration | interventions — Insulin; insulin degludec; Insulin, Short-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afrezza (Technosphere Insulin) + insulin degludec (Experimental): The Afrezza-Degludec group will inhale Afrezza at meals and corrections and will inject insulin degludec once a day for the 17 weeks of the RCT Phase. Dexcom Continuous Glucose Monitoring (CGM) will be provided. The Afrezza-Degludec group will continue to use Afrezza and insulin degludec for an additional 13 weeks in the Extension Phase.
  Interventions: Biological: Afrezza; Biological: insulin degludec
- Usual Care: Insulin delivery with either MDI, a pump without automation, or an AID system and CGM (Active Comparator): The Usual Care group will continue to receive insulin as they did before the study. This could be by multiple daily injections (MDI) or by using an insulin pump with or without automation for the 17 weeks of the randomized controlled trial (RCT) Phase. Participants will continue to use their personal continuous glucose monitor (CGM) as they did before the study. The Usual Care group will then use Afrezza and insulin degludec for 13 weeks in the Extension Phase. Dexcom CGM will be provided during the Extension Phase.
  Interventions: Biological: Rapid-acting Insulin Analog; Biological: Basal Insulin

INTERVENTIONS:
Biological: Afrezza — Pharmaceutical form: powder Route of administration: inhalation
  Other Names: Technosphere Insulin
  Arms: Afrezza (Technosphere Insulin) + insulin degludec
Biological: insulin degludec — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Afrezza (Technosphere Insulin) + insulin degludec
Biological: Rapid-acting Insulin Analog — Pharmaceutical form: clear and colorless solution for injection Route of administration: subcutaneous
  Other Names: any FDA approved Rapid-acting Insulin Analog
  Arms: Usual Care: Insulin delivery with either MDI, a pump without automation, or an AID system and CGM
Biological: Basal Insulin — Pharmaceutical form: clear and colorless solution for injection Route of administration: subcutaneous
  Other Names: any FDA approved Basal Insulin
  Arms: Usual Care: Insulin delivery with either MDI, a pump without automation, or an AID system and CGM

SUMMARY:
INHALE-3 is a Phase 4, randomized controlled trial (RCT) that will randomly assign participants ≥18 years of age with type 1 diabetes (T1D) using multiple daily injections (MDI), an automated insulin delivery (AID) system, or a pump without automation, and continuous glucose monitoring (CGM) 1:1 to an insulin regimen of insulin degludec plus inhaled insulin (Afrezza) and CGM or continuation of usual care. The primary outcome of the RCT is at 17 weeks. The RCT will be followed by a 13-week extension phase in which participants in both groups will use the degludec-inhaled insulin regimen.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent for study participation
* Clinical diagnosis of T1D (per the Investigator)
* Treatment with insulin for at least 6 months prior to the collection of the baseline continuous glucose monitoring (CGM) data
* Same treatment regimen (MDI, an AID system, or an insulin pump without automation) for the 3 months prior to screening

  1. Current (at time of screening) rapid-acting insulin analog (RAA) in use for at least 4 weeks
  2. If AID system used, automated insulin delivery must be active >85% of the time in the 4 weeks prior to screening
  3. If MDI used, participant must be using a long-acting basal insulin plus injecting a RAA bolus for meals, per Investigator
* Total daily insulin dose 20-100 units
* Age ≥ 18 years
* HbA1c <11.0%
* Participant uses real-time CGM (any type of real-time CGM) on a regular basis (at least 70% of the time in the 4 weeks prior to screening)
* No use of inhaled insulin in the 3 months prior to screening
* If female of childbearing potential, willing and able to have pregnancy testing
* Investigator believes that the participant can safely use the study treatment and will follow protocol
* No medical, psychiatric,or other conditions, or medications being taken that in the Investigator's judgement would be a safety concern for participation in the study

  1. This includes considering the potential impact of medical conditions known to be present including cardiovascular, liver, kidney disease, thyroid disease, adrenal disease, malignancies, vision difficulties, active proliferative retinopathy, and other medical conditions; psychiatric conditions including eating disorders; drug or alcohol abuse.

Exclusion Criteria:

* History of recent blood transfusions (within previous 3 months prior to randomization), hemoglobinopathies, (sickle cell trait is not an exclusion), or any other conditions that affect HbA1c measurements
* Recent history of asthma (defined as using any medications to treat within the last year), chronic obstructive pulmonary disease (COPD), or any other clinically important pulmonary disease (e.g., cystic fibrosis or bronchopulmonary dysplasia), or significant congenital or acquired cardiopulmonary disease as judged by the Investigator
* Exposure to any investigational product(s), including drugs or devices, in the 90 days prior to the start of screening
* Any disease other than diabetes or current use (or anticipated use during the study) of any medication that, in the judgment of the Investigator, may impact glucose metabolism
* Current or anticipated acute uses of oral, inhaled or injectable glucocorticoids during the time period of the trial (topical glucocorticoid use is acceptable)
* Use of a non-insulin glucose-lowering medication within 3 months prior to signing informed consent
* Smoking (includes cigarettes, cigars, pipes, marijuana, and vaping devices) within 3 months prior to screening
* Pregnant or lactating, planning to become pregnant during the study, or is a woman of childbearing potential and not on an acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD, or implant); childbearing means that menstruation has started, and the participant is not surgically sterile or greater than 12 months post-menopausal
* No known stage 4/5 renal failure or on dialysis
* Taking Hydroxyurea medication
* An event of severe hypoglycemia, as judged by the Investigator, within the last 90 days prior to screening
* An episode of diabetic ketoacidosis (DKA) diagnosed at a health care facility within the 90 days prior to screening or severe hypoglycemia event within the 90 days prior to screening
* Employed by, or having immediate family members employed by MannKind Corporation or JAEB Center for Health Research, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as Study Investigator, coordinator, etc.); or having a first-degree relative who is directly involved in in conducting the clinical trial
* Have a history or current diagnosis of lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) | 17 weeks
  Change in HbA1c from baseline to 17 weeks (non-inferiority margin 0.4%)

SECONDARY OUTCOMES:
Continuous Glucose Monitoring (CGM) measured percent time with glucose less than 54 mg/dL | 17 weeks
  CGM-measured percent time with glucose <54 mg/dL from baseline to 17 weeks (non-inferiority, margin 0.5%)
Continuous Glucose Monitoring (CGM) measured percent time with glucose less than 70 mg/dL | 17 weeks
  CGM-measured percent time with glucose <70mg/dL from baseline to 17 weeks (non-inferiority, margin 2.0%)
Continuous Glucose Monitoring (CGM) measured daytime (0600-midnight) percent time in range with glucose 70-180 mg/dL | 17 weeks
  CGM-measured daytime (0600-midnight) percent time in range with glucose 70-180 mg/dL from baseline to 17 weeks, for superiority assessment
Mean Continuous Glucose Monitoring (CGM) glucose | 17 weeks
  Mean CGM glucose from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured (24-hours) percent time in range (TIR) with glucose 70-180 mg/dL | 17 weeks
  CGM-measured (24-hours) percent time in range with glucose 70-180 mg/dL from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured percent time with glucose greater than 180 mg/dL | 17 weeks
  CGM-measured percent time with glucose > 180 mg/dL from baseline to 17 weeks, for superiority assessment
Change in glycated hemoglobin (HbA1c) for superiority assessment | 17 weeks
  HbA1c from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured time with glucose greater than 250 mg/dL | 17 weeks
  CGM-measured time with glucose >250 mg/dL from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured time with glucose less than 70 mg/dL | 17 weeks
  CGM-measured time with glucose <70 mg/dL from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured time with glucose less than 54 mg/dL | 17 weeks
  CGM-measured time with glucose <54 mg/dL from baseline to 17 weeks, for superiority assessment
Continuous Glucose Monitoring (CGM) measured coefficient of variation | 17 weeks
  CGM-measured coefficient of variation from baseline to 17 weeks, for superiority assessment
Change in HbA1c less than 7.0% at 17 weeks | 17 weeks
  HbA1c <7.0% at 17 weeks
Change in HbA1c from baseline to 17 weeks, with an improvement of greater than 0.5% | 17 weeks
  HbA1c improvement from baseline to 17 weeks >0.5%
Change in HbA1c from baseline to 17 weeks, with an improvement of greater than 1.0% | 17 weeks
  HbA1c improvement from baseline to 17 weeks >1.0%
Percent time in range (TIR) with glucose 70-140 mg/dL | 17 weeks
  Percent time in range with glucose 70-140 mg/dL
Percent time with glucose greater than 300 mg/dL | 17 weeks
  Percent time with glucose >300 mg/dL
Continuous Glucose Monitoring (CGM) measured prolonged hyperglycemia events | 17 weeks
  CGM-measured prolonged hyperglycemia events
Continuous Glucose Monitoring (CGM) measured hypoglycemia events | 17 weeks
  CGM-measured hypoglycemia events
Standard Deviation (SD) of glucose | 17 weeks
  SD of glucose
"Fasting glucose" by Continuous Glucose Monitoring (CGM) | 17 weeks
  "Fasting glucose" by CGM (defined as closest value to 6 a.m.; assumed, but not verified, with no food during the prior 4-hour period)
Percent time in range (TIR) with glucose 70-180 mg/dL greater than 70% | 17 weeks
  Percent time in range with glucose 70-180 mg/dL >70% at 17 weeks
Percent time in range (TIR) with glucose 70-180 mg/dL improvement from baseline to 17 weeks greater than or equal to 5% | 17 weeks
  Percent time in range with glucose 70-180 mg/dL improvement from baseline to 17 weeks ≥5%
Percent time in range (TIR) with glucose 70-180 mg/dL improvement from baseline to 17 weeks ≥10% | 17 weeks
  Percent time in range with glucose 70-180 mg/dL improvement from baseline to 17 weeks ≥10%
Percent time with glucose less than 70 mg/dL less than 4% | 17 weeks
  Percent time with glucose <70 mg/dL <4% at 17 weeks
Percent time with glucose less than 54 mg/dL less than1% | 17 weeks
  Percent time with glucose <54 mg/dL <1% at 17 weeks
Percent time in range (TIR) 70-180 mg/dL greater than 70% and time less than 54 mg/dL less than 1% | 17 weeks
  Percent time in range 70-180 mg/dL >70% and time <54 mg/dL <1% at 17 weeks
Incidence of severe hypoglycemia events | 30 weeks
  Incidence of severe hypoclycemia events, defined as events requiring assistance of another person due to cognitive impairment to actively administer carbohydrate, glucagon, or other resuscitative actions
Continuous Glucose Monitoring (CGM) measured percent time with glucose less than 54 mg/dL | 30 weeks
  CGM-measured percent time with glucose less than 54 mg/dL
Other serious adverse events, including hospitalizations | 30 weeks
  Other serious adverse events, including hospitalizations
Incidence and severity of treatment-emergent adverse events (TEAEs) | 30 weeks
  Incidence and severity of treatment-emergent adverse events (TEAEs)
Incidence and severity of adverse events of special interest (AESIs) as well as the number of participants with AESIs and number of individual events | 30 weeks
  Incidence and severity of adverse events of special interest (AESIs) as well as the number of participants with AESIs and number of individual events
Change from baseline to 17 weeks in Forced Expiratory Volume in one second (FEV1) | 17 weeks
  Change from baseline to 17 weeks in FEV1
Proportion of participants with Forced Expiratory Volume in one second (FEV1) reduction greater than or equal to 20% | 30 weeks
  Proportions of participants in each group who have experienced ≥20% reduction in FEV1 from baseline to Week 17
Hypoglycemic events from logged blood glucose measurements (BGM): Level 1 events (less than 70 mg/dL) and Level 2 events (less than 54 mg/dL) separately | 30 weeks
  Hypoglycemic events from logged BGM measurements: Level 1 events (<70 mg/dL) and Level 2 events (<54 mg/dL)
Hyperglycemic events from logged blood glucose measurements (BGM) | 30 weeks
  Hyperglycemic events from logged BGM measurements
Continuous Glucose Monitoring (CGM) measured prolonged hyperglycemia events | 30 weeks
  CGM-measured prolonged hyperglycemia events
Continuous Glucose Monitoring (CGM) measured hypoglycemia events (both a safety and efficacy endpoint) | 30 weeks
  CGM-measured hypoglycemia events (both a safety and efficacy endpoint)

OTHER OUTCOMES:
Weight | 17 weeks
  Weight
Post prandial glucose for first meal challenge | 17 weeks
  Post prandial glucose for first meal challenge
Area under the curve (AUC) for first meal challenge | 17 weeks
  Area under the curve (AUC) for first meal challenge
Patient-reported outcome (PRO) questionnaires | 17 weeks
  Type 1 Diabetes Distress Scale (T1-DDS): 28-item validated survey pertaining to distress symptoms related to diabetes (recorded from a scale of 1 to 6).
  Hypoglycemia Confidence Scale (HCS): 9-item validated survey pertaining to situations where hypoglycemia could occur and queries about the participant's level of confidence in those situations (recorded from a scale 1 to 4).
  Insulin Treatment Satisfaction Questionnaire (ITSQ): 22-item survey with a 5-factor structure assessing insulin satisfaction (scores range from 0 to 100).
  Freedom and Flexibility: 6-item non-validated survey pertaining to life experiences impacted by having diabetes (scores range from 6 to 36)
  Insulin Adherence: 1-item non-validated survey pertaining to number of missed boluses in the past week
Change in HbA1c from baseline to 17 weeks, with a worsening of greater than 0.5% | 17 weeks
  Additional binary HbA1c endpoints, HbA1c worsening from baseline to 17 weeks >0.5%
Change in HbA1c from baseline to 17 weeks, with a worsening of greater than 1.0% | 17 weeks
  Additional binary HbA1c endpoints, HbA1c worsening from baseline to 17 weeks >1.0%
Percent time in range (TIR) with glucose 70-180 mg/dL worsening from baseline to 17 weeks greater than or equal to 5% | 17 weeks
  Additional binary CGM endpoints, Percent time in range with glucose 70-180 mg/dL worsening from baseline to 17 weeks ≥5%
Percent time in range (TIR) with glucose 70-180 mg/dL worsening from baseline to 17 weeks greater than or equal to 10% | 17 weeks
  Additional binary CGM endpoints, Percent time in range with glucose 70-180 mg/dL worsening from baseline to 17 weeks ≥10%

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kaiserman, MD, Study Director — Mannkind Corporation; Irl B. Hirsch, MD, Study Chair — University of Washington
Locations (19):
- United States (19):
  - Loma Linda University-Diabetes Treatment Center, Loma Linda, California
  - Sansum Diabetes Research, Santa Barbara, California
  - Barbara Davis Center, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Northwestern University Division of Endocrinology, Metabolism and Molecular Medicine, Chicago, Illinois
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Las Vegas Endocrinology, Henderson, Nevada
  - Endocrine Associate of West Village, PC, Long Island City, New York
  - Mount Sinai Diabetes Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - University of Washington Diabetes Institute, Seattle, Washington
  - Mountain State Diabetes, Parkersburg, West Virginia